CLINICAL TRIAL: NCT00297219
Title: The Effects of Lowering Dialysate Calcium Level on Progression of Coronary Artery Calcification and Bone Histomorphometry: Prospective, Randomized, Controlled Study
Brief Title: Effects of Lowering Dialysate Calcium Level on Progression of Coronary Artery Calcification and Bone Histomorphometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: University of Kentucky (Other); Fresenius Medical Care North America (Industry)
Responsible Party: Ege University, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGE99803466003-2; MO1RR02602NCRR
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: End-Stage Renal Disease; Hemodialysis
Keywords: Hemodialysis; Coronary artery calcification; Adynamic bone disease; Dialysate calcium; Bone mineral density; Bone histomorphometry
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): high dialysate calcium
  Interventions: Drug: high dialysate calcium
- 1 (Active Comparator): low dialysate calcium
  Interventions: Drug: Low dialysate calcium

INTERVENTIONS:
Drug: Low dialysate calcium — 1.25 mmol/L dialysate calcium
  Arms: 1
Drug: high dialysate calcium — 1.75 mmol/L dialysate calcium
  Arms: 2

SUMMARY:
The high rate of cardiovascular complications in the dialysis population cannot be explained by traditional cardiovascular risk factors. One of such factors proposed to contribute to the cardiovascular mortality in dialysis patient population is vascular calcification possibly resulting from disturbances of calcium-phosphate metabolism.

The aim of this study is to assess the effects of treatment with dialysate containing 1.75 or 1.5 mmol/L to 1.25 mmol/L calcium regarding coronary artery calcification and bone histomorphometry in hemodialysis patients.

DETAILED DESCRIPTION:
Sample size calculations were based on previously reported changes in coronary artery calcification scores in hemodialysis patients during time (90% power with a two-sided, alpha error rate of 5%). Four hundred fifty-seven hemodialysis patients, taking drop-out rate into consideration, will be enrolled in this prospective-controlled study.The cases already being treated with calcium-based phosphate binder and dialysate containing 1.75 or 1.5 mmol/L calcium will be enrolled from eight hemodialysis centers.The cases will be randomized to two arms:

1. Dialysate containing 1.25 mmol/L calcium + calcium-based phosphate binder group: Dialysate calcium will be reduced from 1.75 or 1.5 mmol/L to 1.25 mmol/L in this group. Patients will use calcium-based phosphate binder according to phosphate level.
2. Dialysate containing 1.75 mmol/L calcium + calcium-based phosphate binder group (Control group): Dialysate calcium will remain or switched to 1.75 mmol/L and patients will be on calcium-based phosphate binder.

The study will last for 18 months.Coronary artery calcification (Multi-slice CT), bone histomorphometry, and bone mineral density will be assessed in the beginning and at the end of the study. Coronary artery calcification and bone mineral density will be measured in all patients; bone histomorphometry will be assessed in 150 patients, 75 from each group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* On maintenance bicarbonate hemodialysis scheduled thrice weekly, at least 12 hours/week
* To be treated with a dialysate containing 1.75 or 1.5 mmol/L calcium
* Willingness to participate in the study with a written informed consent

Exclusion Criteria:

* To be scheduled for living donor renal transplantation
* To have serious life-limiting co-morbid situations, namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease
* Pregnancy or lactating
* To be unable to give informed consent because of mental incompetence or a psychiatric disorder
* To be on vitamin D treatment within six months of randomization or having iPTH values over target levels (>300 pg/mL)
* Hypercalcemia (Ca >10.5 mg/dl) with use of dialysate containing 1.75 or 1.5 mmol/L calcium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Progression of coronary artery calcification scores | eighteen months
Changes in bone histomorphometry analysis | eighteen months
Changes in bone mineral density | eighteen months

SECONDARY OUTCOMES:
Changes in intact PTH levels | eighteen months
effects of dialysate with or without glucose (e.g intradialytic hypoglycemia and hypotension, arrythmia-by Holter ECG- and changes in HbA1c, insulin) | eighteen months

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, MD, Principal Investigator — Ege University School of Medicine Nephrology Department
Locations (3):
- University of Kentucky Medical Center, Lexington, Kentucky, United States
- Turkey (Türkiye) (2):
  - FMC Clinics, Bornova, İzmir
  - Ege University School of Medicine, Bornova-Izmir